CLINICAL TRIAL: NCT05369689
Title: Stereotactic Radiosurgery Prognosis Assessment for Spinal Tumors Based on Radiomics
Status: Not yet recruiting | Type: Observational
Sponsor: Zhuang Hongqing (Other)
Responsible Party: Sponsor-Investigator, Zhuang Hongqing, Associate department chairman of radiotherapy, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Other Study IDs: SBRTradiomics
Record Dates: First submitted 2022-05-07; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Stereotactic Radiosurgery; Spinal Tumor; Radiomics; Prognosis
MeSH Terms: conditions — Spinal Cord Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- spinal tumors, CT, MRI, PET-CT stereotactic radiosurgery: Patients who had spinal tumors and completed the CT, MRI or PET-CT examination before and after stereotactic radiosurgery.
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — As this is a prognosis evaluation study, there are no interventions.

SUMMARY:
This study aims to assess multimodal Radiomics-based prediction model for prognostic prediction in spinal tumors.

DETAILED DESCRIPTION:
Sensitivity for prediction recurrence and survival of currently available prognostic scores is limited. This study proposes to establish a multimodal radiomics model for identifying tumor recurrence and prognostic prediction of spinal tumors. The study will investigate the relationship between the radiomics and the tumor microenvironment. The study includes the construction of multimodal radiomics-based prediction model and the validation of the prediction model.

ELIGIBILITY:
Inclusion Criteria:

A diagnosis of spinal tumors for which SBRT is appropriate Karnofsky Performance Status >60 Life expectancy of at least 3 months No contraindication to undergoing MR imaging Age >18 Complete the CT MRI or PET-CT examination before and after treatment Accept stereotactic radiosurgery

Exclusion Criteria:

Subjects unable to undergo MRI (includes non-MRI compatible material or devices and severe claustrophobia) Subjects with prior procedural intervention to the involved vertebral body that would result in artifact (kyphoplasty, screw and/or rod placement); minimally invasive surgery without instrumentation of the involved vertebral body and instrumentation immediately above or below the index lesion is allowed.

Subjects with spinal cord compression; minimally invasive "separation" surgery to first resect the epidural component is allowed Pregnant or breast-feeding women Allergy to standard IV contrast agents used in MRI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had spinal tumors and completed CT, MRI, PET-CT examination before and after stereotactic radiosurgery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 1 years
  progression-free survival

SECONDARY OUTCOMES:
Overall survival (OS) | 1 years
  defined as the time from the beginning of diagnosis of spinal tumors to the death with any causes
ORR | 3 months
  objective response rate
DCR | 3 months
  disease control rate
Recurrence free survival (RFS) | 1 year
  defined as time between randomization and the time of any recurrence of ipsilateral chest, breast, regional lymph node recurrence, distant metastases, or death occurred

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology Cancer Center, Peking University Third Hospital 49# North Garden Rd.,Haidian Dist., Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No